CLINICAL TRIAL: NCT00982631
Title: A Phase Ib Study of Combination of Temsirolimus (Torisel®) and Pegylated Liposomal Doxorubicin (PLD, Doxil®/ Caelyx®) in Advanced or Recurrent Breast, Endometrial and Ovarian Cancer
Brief Title: A Study of Combination of Temsirolimus (Torisel®) and Pegylated Liposomal Doxorubicin (PLD, Doxil®/Caelyx®) in Advanced or Recurrent Breast, Endometrial and Ovarian Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCNONCO200902
Record Dates: First submitted 2009-09-17; First posted 2009-09-23 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Advanced/Recurrent Breast Cancer; Endometrial Cancer; Ovarian Cancer
Keywords: temsirolimus (Torisel®); pegylated liposomal doxorubicin (PLD, Doxil®/ Caelyx®)
MeSH Terms: conditions — Breast Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- temsirolimus/PLD (Experimental): temsirolimus (Torisel) with pegylated liposomal doxorubicin (PLD,Doxil,Caelyx);a dose escalating study in a 3+3 design
  Interventions: Drug: Temsirolimus/PLD

INTERVENTIONS:
Drug: Temsirolimus/PLD — This is a dose escalation study. Patients will start with temsirolimus iv once weekly. After 2 weeks, PLD therapy is added. From then on, PLD is repeated every 4 weeks. One cycle is 28 days. The DLT period is also defined within the first 28 days of combination therapy (thus the first 6 weeks of study participation). The first dose level (DL) is DL 1. Depending on toxicity, intermediate dose levels can be added. If no MTD is found in the sixth cohort, this dose level will be considered as the recommended dose (RD), being the optimal dose for both drugs in this combination. At the MTD dose level, the dose level will be expanded to a total of 12 patients.

SUMMARY:
A study to examine the combination of temsirolimus and Caelyx® (chemotherapeutic) in advanced or recurrent breast, endometrial and ovarian cancer.

DETAILED DESCRIPTION:
To assess the maximum tolerated dose (MTD) and recommended phase II dose of the combination of temsirolimus and Caelyx® in patients with advanced or therapy refractory breast cancer, endometrial cancer, or ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven advanced breast cancer, endometrial cancer or ovarian cancer, who are refractory to standard therapies or for whom no standard therapy exists.
* Age ≥ 18 years
* Patients who have an ECOG status of 0 or 1
* Patients who have a life expectancy of at least 12 weeks
* Negative pregnancy test for female patients of childbearing potential
* Signed informed consent

Exclusion Criteria:

* Adequate bone marrow: neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L and haemoglobin ≥ 5.0 mmol/l
* Adequate renal function: GFR ≥ 60 ml/min
* Adequate liver function: ALT and AST < 2.5 x ULN, total bilirubin ≤ 1x ULN
* Fasting level of total cholesterol of no more than 350 mg/dL (9.1 mmol/L) and triglyceride level of no more than 400 mg/L (4.5 mmol/L)
* Left ventricular ejection fraction (LVEF) < 50%
* History of serious cardiac disease
* Active clinically serious bacterial, viral or fungal infections (> grade 2).
* Known history of human immunodeficiency virus (HIV) infection or chronic hepatitis B or C.
* Clinically symptomatic brain or meningeal metastasis. Patients with seizure disorders requiring medication (such as steroids or antiepileptics). Concomitant treatment with strong CYP3A4 inductors (such as rifampicin, St. John´s Wort) or CYP3A4 inhibitors (such as ketoconazole, voriconazole, itraconazole, diltiazem, verapamil, erythromycin) within 2 weeks prior to start.
* Moderate or weak CYP3A4 modifiers should be used concomitantly only after careful assessment of risk-benefit ratio. Concomitant use of carbamazepine, phenobarbital, phenytoin or chronic use of dexamethasone is not allowed. (Table 1)
* Other concomitant anti-cancer therapy (except steroids)
* Concomitant use of streptozocin, mercaptopurine.
* Previous treatment with one of the study drugs.
* Previous treatment with other mTOR inhibitors
* Prior investigational therapy/agents within 4 weeks of start, in case of bevacizumab at least 60 days between bevacizumab discontinuation and first dosing of temsirolimus.
* Surgical treatment or radiation therapy in the past 4 weeks. Palliative radiotherapy at focal sites on the extremities is allowed, also within 4 weeks before start
* Unresolved toxicity CTC ≥ grade 2 from previous anti-cancer therapy except alopecia.
* Known or suspected allergy to any investigational agent or any agent given in association with this trial.
* Substance abuse, medical, psychological or social conditions that may interfere with the patients participation in the study or evaluation of the study results
* Any condition that is unstable or which could jeopardize the safety of patient and his compliance in the study.
* Antracyclines: > 450 mg/m2 doxorubicin or and > 600 mg/m2 epirubicin
* Medications known to have dysrhythmic potential is not permitted (ie, terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide)
* Usage of coumarin-derivate anticoagulants. Low molecular weight heparin is permitted and advised

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
MTD, pharmacokinetic parameters | 2 years

SECONDARY OUTCOMES:
Effectiveness: objective response rate, time to progression | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: C.M.L. van Herpen, MD, Phd, Principal Investigator — UMCN st Radboud
Locations (1):
- University Medical Center Nijmegen st Radboud, Nijmegen, Gelderland, Netherlands